CLINICAL TRIAL: NCT06355674
Title: Effect of Breastfeeding Education Given to Adolescent Mothers With Lactation Simulation Model on Maternal Breastfeeding Self-Efficacy, Maternal Infant Attachment, and Infant Anthropometric Measurements
Brief Title: Adolescent Mother and Breastfeeding Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adiyaman University (Other)
Responsible Party: Principal Investigator, Maksude YILDIRIM, Assistant Professor, Adiyaman University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: HRÜ/23.21.12
Record Dates: First submitted 2024-03-23; First posted 2024-04-09 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Adolescent Mother

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breastfeeding education group (Experimental): Adolescent mothers included in the breastfeeding education group will receive practical breastfeeding training using the lactation simulation model and newborn baby mannequin for 1.5-2 hours conducted by the researchers.
  One week and one month after postnatal day 7, the "Postnatal Breastfeeding Self-Efficacy Scale - Short Form" and the "Maternal-Infant Attachment Scale" will be administered again to mothers in both groups.
  Anthropometric measurements of all babies will be repeated and recorded at the end of the 1st, 2nd, 3rd, and 4th weeks following postnatal day 7.
  After the completion of the study, adolescent mothers in the control group who request it will receive breastfeeding education using the lactation simulation model provided by the researchers.
  Interventions: Behavioral: Breastfeeding education provided with Lactation Simulation Model
- Control group (No Intervention): Adolescent mothers in the control group will continue with routine breastfeeding and follow-up at the family health center.
  One week and one month after postnatal day 7, the "Postnatal Breastfeeding Self-Efficacy Scale - Short Form" and the "Maternal-Infant Attachment Scale" will be administered again to mothers in both groups.
  Anthropometric measurements of all babies will be repeated and recorded at the end of the 1st, 2nd, 3rd, and 4th weeks following postnatal day 7.
  After the completion of the study, adolescent mothers in the control group who request it will receive breastfeeding education using the lactation simulation model provided by the researchers.

INTERVENTIONS:
Behavioral: Breastfeeding education provided with Lactation Simulation Model — The Lactation Simulation Model (LSM) is a high-fidelity simulator designed for interactive education, which educators can utilize for practical and wearable breastfeeding training. It is wearable like a shirt and is secured onto the chest by passing it over the shoulders and fastening it with a safety belt from the back. This allows the safety belt to be adjusted according to different body types and weights.
  Arms: Breastfeeding education group

SUMMARY:
In low-income and developing countries, 30% of adolescents marry before the age of 18, and 14% marry before the age of 15. Additionally, adolescents between the ages of 15 and 19 are often coerced into marriage or sexual relationships with partners older than themselves. 10% of adolescents under the age of 15 in the world are forced to have sexual intercourse and as a result, unwanted teenage pregnancies occur. In high-income countries like Latin America, there is a high prevalence of adolescent non-marital pregnancies. When considering the fertility, health, and social outcomes of adolescence, it emerges as a significant issue. Adolescent motherhood carries numerous adverse effects from both demographic and social perspectives.

In pregnancies occurring during adolescence, both maternal and infant mortality rates are two to three times higher compared to pregnancies at later ages. Many infant and child deaths occur due to preventable causes. Breastfeeding is a significant factor in reducing infant and child mortality. Since infants born to adolescent mothers are at higher risk of death and illness, breastfeeding these infants becomes even more important. However, one of the significant challenges adolescent mothers face during the postpartum period is initiating and maintaining lactation. Research has shown that maternal age plays a significant role in initiating and sustaining breastfeeding, with a strong positive correlation between maternal age and duration of breastfeeding. This study was designed as a randomized controlled trial to examine the effect of breastfeeding education provided to adolescent mothers on maternal breastfeeding self-efficacy, mother-infant attachment, and infant anthropometric measurements.

ELIGIBILITY:
Inclusion Criteria:

* Giving birth vaginally between the 37th and 40th gestational weeks,
* Being under 18 years of age,
* Primigravida,
* Not having any systemic/chronic diseases,
* Willing to breastfeed,
* Having received breastfeeding counseling provided by the hospital,
* Being able to speak Turkish, and
* Adolescent mothers in the postnatal 1st and 2nd weeks will be included in the study.

Exclusion Criteria:

* Mothers giving birth before the 37th gestational week or after the 40th gestational week,
* Those with barriers hindering effective communication,
* Those unable to speak Turkish,
* Mothers who have not received breastfeeding counseling from the hospital,
* Non-breastfeeding mothers,
* Those experiencing interruptions in breastfeeding due to seasonal work or any other reason,
* Those supplementing breastfeeding with formula,
* Adolescent mothers who discontinue breastfeeding education provided through LSM will be excluded from the study.

Ages: 12 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2024-02-12 (Actual); Primary Completion 2024-07-17 (Actual); Study Completion 2024-07-17 (Actual)

PRIMARY OUTCOMES:
Postnatal Breastfeeding Self-Efficacy Scale-Short Form | 4 months
  The short form of the scale consists of a total of 14 items and is a 5-point Likert scale. Scores on the scale can range from 14 to 70 points. A higher score indicates higher maternal breastfeeding self-efficacy.
Maternal-Infant Attachment Scale | 4 months
  The scale consists of a total of eight items rated on a four-point Likert scale. An increase in scores on the scale indicates an improvement in mother-infant attachment.

CONTACTS AND LOCATIONS:
Locations (1):
- Harran University, Sanliurfa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No